CLINICAL TRIAL: NCT03944707
Title: A Randomized, Subject- and Investigator-blinded, Placebo-controlled Study to Assess the Efficacy and Safety of LOU064 in Patients With Inadequately Controlled Asthma
Brief Title: Study of Efficacy and Safety of LOU064 in Inadequately Controlled Asthma Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Company decision
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLOU064D12201; 2018-003609-24 (EudraCT Number)
Record Dates: First submitted 2019-05-02; First posted 2019-05-09 (Actual); Results first posted 2021-04-27 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: Asthma
Keywords: asthma; LOU064
MeSH Terms: conditions — Asthma | interventions — remibrutinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LOU064 (Experimental): LOU064 100 mg once daily orally
  Interventions: Drug: LOU064 100 mg
- Placebo (Placebo Comparator): Placebo once daily orally
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LOU064 100 mg — LOU064 100 mg once daily orally administered as two 50 mg capsules
  Arms: LOU064
Drug: Placebo — Placebo once daily administered orally as capsules
  Arms: Placebo

SUMMARY:
This was a proof-of-concept study to evaluate the efficacy of LOU064 in patients with inadequately controlled asthma. All subjects were randomized with 3:2 ratio to receive LOU064 100 mg once daily or LOU064 matching placebo for 12 weeks with standard background therapy of budesonide 80 µg/formoterol 4.5 µg two inhalations twice a day (b.i.d).

DETAILED DESCRIPTION:
This was a non-confirmatory, multi-center, randomized, placebo-controlled, subject- and investigator-blinded, parallel-group study to evaluate the efficacy and safety of LOU064 in patients with inadequately controlled asthma who were on a standardized background therapy of inhaled corticosteroid plus long acting beta-2 agonist (ICS/LABA).

The study included:

* a Screening period of up to 2 weeks to assess eligibility.
* a Run-in period of minimum 3 weeks and maximum 5 weeks where patients discontinued their current asthma therapy and were placed on budesonide 80 μg/formoterol 4.5 μg delivered by dry powder inhaler, two inhalations twice a day (b.i.d).
* a Treatment period of 12 weeks. All subjects were randomized 3:2 to receive LOU064 100 mg once daily or placebo for 12 weeks with standard background therapy of budesonide 80 μg/formoterol 4.5 μg, two inhalations b.i.d.
* a Follow-up period of 3 weeks following the last dose of study drug. Results from the interim analysis did not provide sufficient evidence of efficacy of LOU064 in inadequately controlled asthma and the sponsor decided to terminate early the study in April 2020. The median duration of exposure (12.0 weeks for LOU064 and 11.7 weeks for placebo) was close to the treatment target, as most of the subjects had completed treatment when the study was terminated.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adult patients aged ≥ 18 to ≤ 70 years at screening.
* Patients must weigh at least 40 kg to participate in the study, and must have a body mass index (BMI) <35 kg/m2. BMI = Body weight (kg) / [Height (m)]2 at screening
* Patients with a physician-diagnosed history of asthma (according to GINA 2018) for a period of at least 6 months prior to screening.
* Patients who have been treated with:

  * Medium or high dose inhaled corticosteroids (ICS), or
  * ICS plus long-acting beta agonist (LABA), or
  * ICS plus leukotriene receptor antagonist (LTRA), or
  * ICS plus long-acting beta agonist (LABA) and long lasting muscarinic antagonist (LAMA) for at least 1 month prior to screening and on the same doses of the above mentioned medications over at least 2 weeks prior to start of the run-in period.
* Post-bronchodilator reversibility of FEV1 ≥ 12% and ≥ 200 mL at screening. If reversibility is not demonstrated at screening, then two additional attempts are permitted (one at the run-in visit and the last one during the run-in period between the run-in visit and baseline visit if needed)
* Spirometry with pre-bronchodilator FEV1 ≥ 40% of predicted (at screening and baseline) and ≤ 85% of predicted at the baseline visit.
* ACQ-5 score ≥ 1.5 at baseline visit
* ≥ 80% compliance with peak expiratory flow measurement and recording of symptoms in the eDiary during the run-in period.

Exclusion Criteria:

* Patients who have had an asthma exacerbation requiring systemic corticosteroids, hospitalization, or emergency room visit within 6 weeks prior to screening or during the screening period.
* Patients who have smoked or inhaled any substance other than asthma medications within the 6 month period prior to screening, or who have a smoking history of greater than 10 pack years (e.g. 10 pack years = 1 pack/day x 10 years or ½ pack/day x 20 years, etc.).
* History of life-threatening asthma event such as significant hypercarbia (pCO2 > 45 mmHg), endotracheal intubation, non-invasive positive pressure ventilation (NIPPV), respiratory arrest, or seizure as a result of asthma.
* Patients with chronic lung diseases other than asthma, including (but not limited to) chronic obstructive pulmonary disease, clinically significant bronchiectasis, sarcoidosis, interstitial lung disease, cystic fibrosis, Churg-Strauss syndrome, allergic broncho-pulmonary aspergillosis, or clinically significant chronic lung diseases related to a history of tuberculosis or asbestosis.
* History or current diagnosis of ECG abnormalities indicating significant risk of safety for subjects participating in the study such as:

  * Concomitant clinically significant cardiac arrhythmias, e.g. sustained ventricular tachycardia, and clinically significant second or third degree AV block without a pacemaker
  * History of familial long QT syndrome or known family history of Torsades de Pointes
  * Resting heart rate (physical exam or 12 lead ECG) < 50 bpm at screening
  * Resting QTcF ≥ 450 msec (male) or ≥ 460 msec (female) at screening or inability to determine the QTcF interval
  * Use of agents known to prolong the QT interval unless they can be permanently discontinued for the duration of study
* At screening and/or run-in period, any severe, progressive or uncontrolled, acute or chronic, medical or psychiatric condition, or other factors such as abnormal vital signs, ECG or physical findings, or clinically relevant abnormal laboratory values, that in the judgment of the investigator may increase the risk associated with study participation/treatment or may interfere with interpretation of study results, and thus would make the patient inappropriate for entry into or continuing the study.
* Major surgery within 8 weeks prior to screening or surgery planned prior to end of study.
* History of live attenuated vaccine within 6 weeks prior to randomization or requirement to receive vaccinations at any time during the study.
* Hematology parameters at screening:

  * Hemoglobin: < 10 g/dl
  * Platelets: < 100 000/mm3
  * White blood cells: < 3 000/mm3
  * Neutrophils: < 1 500/mm3
* Significant bleeding risk or coagulation disorders.
* History of gastrointestinal bleeding, e.g. in association with use of Nonsteroidal Anti-Inflammatory Drug (NSAID).
* Requirement for anti-platelet or anticoagulant medication (e.g., warfarin, or clopidogrel or Novel Oral Anti-Coagulant (NOAC)) other than acetylsalicylic acid (up to 100 mg/d).
* History or presence of thrombotic or thromboembolic event, or increased risk for thrombotic or thromboembolic event.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2019-07-18 (Actual); Primary Completion 2020-04-27 (Actual); Study Completion 2020-04-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (16):
- United States (4):
  - Novartis Investigative Site, Denver, Colorado
  - Novartis Investigative Site, North Dartmouth, Massachusetts
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Raleigh, North Carolina
- Argentina (2):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Rosario, Santa Fe Province
- Germany (4):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanover
- Poland (4):
  - Novartis Investigative Site, Biaystok, Poland
  - Novartis Investigative Site, Grudziądz
  - Novartis Investigative Site, Krakow
  - Novartis Investigative Site, Poznan
- Russia (2):
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Ulyanovsk

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.

REFERENCES:
- See also: A Plain Language Trial Summary is available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=810

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in 19 investigative sites in 5 countries.
Pre-assignment Details: After the screening, participants went through a Run-in period of 3-5 weeks where they discontinued their current asthma therapy and were placed on budesonide 80 μg/formoterol 4.5 μg delivered by dry powder inhaler. Afterwards, patients were randomized in 3:2 ratio to receive LOU064 or placebo and continued to use the budesonide/formoterol inhaler.
Period: Overall Study
Arm/Group | LOU064 | Placebo
Started | 47 | 29
PK Analysis Set (All subjects with at least one available valid pharmacokinetics (PK) concentration measurement, who received any study drug and with no protocol deviations that affected PK data.) | 33 | 0
PD Analysis Set (All subjects with available pharmacodynamics (PD) data and no protocol deviations with relevant impact on PD data. A subject with available PD data was a subject with at least one on-treatment spirometry assessment or with PD diary data for at least 14 days.) | 47 | 29
Completed | 35 | 19
Not Completed | 12 | 10
Not completed — Adverse Event | 0 | 2
Not completed — Study terminated by sponsor | 12 | 7
Not completed — Subject decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LOU064 | Placebo | Total
Number analyzed (Participants) | 47 | 29 | 76
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.2 (10.96) | 53.2 (10.40) | 50.7 (10.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 22 | 50
  Male | 19 | 7 | 26
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 42 | 27 | 69
  Black | 4 | 2 | 6
  Asian | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Pre-dose FEV1 at Week 12
Description: FEV1 (forced expiratory volume in one second) is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation, measured through spirometry testing. Pre-dose FEV1 is defined as average of the two FEV1 measurements taken 45 min and 15 min pre-dose.
  The baseline pre-dose FEV1 is defined as the average of the FEV1 measurements performed 45 min and 15 min prior to dosing on Day 1.
  A positive change from baseline in pre-dose FEV1 is considered a favorable outcome.
  Change from baseline in pre-dose FEV1 was analyzed using a Bayesian model for repeated measures, adjusting for effects of treatment*visit interaction and baseline pre-dose FEV1. A weakly informative prior was considered for the placebo response.
Time Frame: Baseline, Week 12
Population: PD analysis set including participants with a valid measurement for the outcome measure.
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | LOU064 | Placebo
Number analyzed (Participants) | 32 | 20
liters | 0.105 (0.0494) | 0.075 (0.0497)
Statistical Analysis 1: Comparison: LOU064 vs Placebo; Test type: Superiority; p = 0.6643, Bayesian model for repeated measures — Probability LOU064 better than placebo; Mean Difference (Net) = 0.030, 80% CI 2-sided [-0.060 to 0.119], Standard Deviation 0.0698 — Posterior mean difference (LOU064 - placebo) and 80% credible interval are presented

2. Secondary Outcome: Maximum Observed Blood Concentrations (Cmax) of LOU064 at Steady State
Description: Pharmacokinetic (PK) parameters were calculated based on LOU064 blood concentrations determined by a validated liquid chromatography and tandem mass spectrometry (LC-MS/MS) method with a lower limit of quantification of 1 ng/mL. Cmax was determined using non-compartmental methods.
Time Frame: pre-dose, 0.5, 1, 2, 3 and 4 hours after dosing on Days 15 and 85
Population: PK analysis set including participants with a valid measurement for the outcome measure.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | LOU064 | Placebo
Number analyzed (Participants) | 33 | 0
ng/mL
  Day 15: number analyzed (Participants) | 32 | 0
  Day 15 | 239 (152) |
  Day 85: number analyzed (Participants) | 22 | 0
  Day 85 | 222 (142) |

3. Secondary Outcome: Time to Reach Maximum Blood Concentrations (Tmax) of LOU064 at Steady State
Description: PK parameters were calculated based on LOU064 blood concentrations determined by a validated LC-MS/MS method with a lower limit of quantification of 1 ng/mL. Tmax was determined using non-compartmental methods.
Time Frame: pre-dose, 0.5, 1, 2, 3 and 4 hours after dosing on Days 15 and 85
Population: PK analysis set including participants with a valid measurement for the outcome measure.
Measure: Median (Full Range); unit: hours (hr)
Arm/Group | LOU064 | Placebo
Number analyzed (Participants) | 33 | 0
hours (hr)
  Day 15: number analyzed (Participants) | 32 | 0
  Day 15 | 1.00 [0.483 to 2.00] |
  Day 85: number analyzed (Participants) | 22 | 0
  Day 85 | 1.00 [0.500 to 3.00] |

4. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero to 24 Hours (AUC0-24h) of LOU064 at Steady State
Description: PK parameters were calculated based on LOU064 blood concentrations determined by a validated LC-MS/MS method with a lower limit of quantification of 1 ng/mL. AUC0-24h was determined using non-compartmental methods. The linear trapezoidal rule was used for AUC0-24h calculation.
Time Frame: pre-dose, 0.5, 1, 2, 3 and 4 hours after dosing on Days 15 and 85
Population: PK analysis set including participants with a valid measurement for the outcome measure.
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | LOU064 | Placebo
Number analyzed (Participants) | 33 | 0
hr*ng/mL
  Day 15: number analyzed (Participants) | 21 | 0
  Day 15 | 471 (285) |
  Day 85: number analyzed (Participants) | 16 | 0
  Day 85 | 517 (342) |

5. Secondary Outcome: Change From Baseline in Asthma Symptom Questionnaire-5 Score (ACQ-5) at Week 12
Description: The ACQ-5 is a five-item, self-completed questionnaire, which is used as a measure of asthma control of a participant. Patients were asked to recall how their asthma had been during the previous week and to respond to the symptom questions on a 7-point scale (0=no impairment, 6=maximum impairment). The questions are equally weighted and the overall ACQ-5 score is the mean of all 5 questions, therefore between 0 (totally controlled) and 6 (severely uncontrolled).
  The baseline values of ACQ-5 were collected at the baseline visit. A negative change from baseline in ACQ-5 is considered a favorable outcome. Change from baseline in ACQ-5 score was analyzed using a Bayesian model for repeated measures, adjusting for effects of treatment*visit interaction and baseline ACQ-5 score. Non-informative priors were considered.
Time Frame: Baseline, Week 12
Population: PD analysis set including participants with a valid measurement for the outcome measure.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | LOU064 | Placebo
Number analyzed (Participants) | 33 | 20
score on scale | -0.95 (0.133) | -0.86 (0.164)
Statistical Analysis 1: Comparison: LOU064 vs Placebo; Test type: Superiority; p = 0.6609, Bayesian model for repeated measures — Probability LOU064 better than placebo; Median Difference (Net) = -0.09, 80% CI 2-sided [-0.35 to 0.18], Standard Deviation 0.210 — Posterior mean difference (LOU064 - placebo) and 80% credible interval are presented

6. Secondary Outcome: Change From Baseline in Mean Morning and Mean Evening Peak Expiratory Flow (PEF)
Description: PEF (Peak Expiratory Flow) is a person's maximum speed of expiration. All participants were instructed to record PEF twice daily before taking any medication using an electronic peak expiratory flow device (ePEF), once in the morning and once approximately 12 h later in the evening at home. At each timepoint, the participant was instructed to perform 3 consecutive manoeuvres within 10 minutes. These PEF values were captured in the e-PEF/diary. For each day the best value in the morning and in the evening were considered and mean values on 4-week intervals were derived.
  The baseline values of PEF were the mean values in the run-in period. A positive change from baseline in PEF is considered a favorable outcome. Change from baseline in mean morning and mean evening PEF were analyzed using a Bayesian model for repeated measures, adjusting for effects of treatment*weeks interaction and baseline PEF values. Non-informative priors were considered.
Time Frame: Baseline, Weeks 9-12
Population: PD analysis set including participants with a valid measurement for the outcome measure.
Measure: Mean (Standard Deviation); unit: liters/minute
Arm/Group | LOU064 | Placebo
Number analyzed (Participants) | 47 | 29
liters/minute
  Change from baseline in mean morning PEF: number analyzed (Participants) | 29 | 18
  Change from baseline in mean morning PEF | -2.4 (4.30) | -2.6 (5.59)
  Change from baseline in mean evening PEF: number analyzed (Participants) | 28 | 18
  Change from baseline in mean evening PEF | -9.7 (5.58) | -6.3 (7.23)
Statistical Analysis 1: Comparison: LOU064 vs Placebo; Change from baseline in mean morning PEF; Test type: Superiority; p = 0.5107, Bayesian model for repeated measures — Probability LOU064 better than placebo; Mean Difference (Net) = 0.1, 80% CI 2-sided [-9.0 to 9.1], Standard Deviation 7.13 — Posterior mean difference (LOU064 - placebo) and 80% credible interval are presented
Statistical Analysis 2: Comparison: LOU064 vs Placebo; Change from baseline in mean evening PEF; Test type: Superiority; p = 0.3611, Bayesian model for repeated measures — Probability LOU064 better than placebo; Mean Difference (Net) = -3.4, 80% CI 2-sided [-15.2 to 8.1], Standard Deviation 9.15 — Posterior mean difference (LOU064 - placebo) and 80% credible interval are presented

7. Secondary Outcome: Change From Baseline in Number of Puffs of SABA Taken Per Day During the Treatment Period
Description: Participants were given a short acting β2-agonist (SABA; salbutamol, known also as albuterol) to use as rescue medication throughout the study along with an electronic diary (eDiary) to record rescue medication use. Participants recorded in the eDiary, once in the morning and once in the evening, the use of rescue medication (number of puffs of SABA taken in the previous 12 hours). The total number of puffs of SABA taken per day was calculated and the mean daily use of puffs of SABA over 12 weeks was derived.
  The baseline values of number of puffs of SABA taken per day were defined as the average from all non-missing records taken during the run-in period. A negative change from baseline is considered a favorable outcome.
  Change from baseline in number of puffs of SABA taken per day was analyzed using a Bayesian model, adjusting for effects of baseline SABA use, baseline FEV1, baseline asthma daytime symptom score and treatment. Non-informative priors were considered.
Time Frame: Baseline, 12 weeks
Population: PD analysis set including participants with a valid measurement for the outcome measure.
Measure: Mean (Standard Deviation); unit: puffs of SABA
Arm/Group | LOU064 | Placebo
Number analyzed (Participants) | 41 | 26
puffs of SABA | -0.192 (0.0946) | -0.059 (0.1224)
Statistical Analysis 1: Comparison: LOU064 vs Placebo; Test type: Superiority; p = 0.8022, Bayesian model — Probability LOU064 better than placebo; Mean Difference (Net) = -0.133, 80% CI 2-sided [-0.336 to 0.071], Standard Deviation 0.1588 — Posterior mean difference (LOU064 - placebo) and 80% credible interval are presented

8. Secondary Outcome: Change From Baseline in Daytime and Nighttime Asthma Symptom Score
Description: Participants recorded asthma symptoms twice daily in the eDiary. Daytime asthma symptoms were assessed before bed and nighttime symptoms on awakening.
  * Daytime asthma symptom score included 4 questions. Overall score (0 to 6) was calculated as the average of the 4 questions with higher values indicating more asthma symptoms.
  * Nighttime asthma symptom score included 2 questions. Overall score (0 to 3.5) was calculated as the average of the 2 questions with higher values indicating more asthma symptoms.
  Mean values of both scores were calculated over 4-week intervals during the treatment period.
  The baseline values of both asthma symptoms scores were defined as the average score during the run-in period. A negative change from baseline is a favorable outcome.
  Change from baseline in daytime and nighttime asthma symptom score were analyzed using a Bayesian model for repeated measures, adjusting for effects of treatment*weeks and baseline scores. Non-informative priors were considered.
Time Frame: Baseline, Weeks 9-12
Population: PD analysis set including participants with a valid measurement for the outcome measure.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | LOU064 | Placebo
Number analyzed (Participants) | 47 | 29
score on scale
  Change from baseline in daytime asthma symptom score: number analyzed (Participants) | 34 | 20
  Change from baseline in daytime asthma symptom score | -0.225 (0.0962) | -0.175 (0.1237)
  Change from baseline in nighttime asthma symptom score: number analyzed (Participants) | 34 | 20
  Change from baseline in nighttime asthma symptom score | -0.120 (0.0488) | -0.195 (0.0651)
Statistical Analysis 1: Comparison: LOU064 vs Placebo; Change from baseline in daytime asthma symptom score; Test type: Superiority; p = 0.6312, Bayesian model for repeated measures — Probability LOU064 better than placebo; Mean Difference (Net) = -0.050, 80% CI 2-sided [-0.251 to 0.149], Standard Deviation 0.1573 — Posterior mean difference (LOU064 - placebo) and 80% credible interval are presented
Statistical Analysis 2: Comparison: LOU064 vs Placebo; Change from baseline in nighttime asthma symptom score; Test type: Superiority; p = 0.1752, Bayesian model for repeated measures — Probability LOU064 better than placebo; Mean Difference (Net) = 0.075, 80% CI 2-sided [-0.028 to 0.180], Standard Deviation 0.0819 — Posterior mean difference (LOU064 - placebo) and 80% credible interval are presented

ADVERSE EVENTS:
Time Frame: From first dose of study treatment until last dose of study treatment plus 30 days post treatment, up to Day 115.
Description: Any sign or symptom that occurs during the study treatment plus 30 days post treatment.
Arm/Group | LOU064 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/29
Other Adverse Events (participants affected / at risk) | 8/47 | 10/29
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LOU064 (N=47) | Placebo (N=29)
Nasopharyngitis (Infections and infestations) | 4 | 6
Upper respiratory tract infection (Infections and infestations) | 4 | 4
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. Novartis does not prohibit any investigator from publishing. Any publications from a single site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-03-18): https://cdn.clinicaltrials.gov/large-docs/07/NCT03944707/Prot_001.pdf
  • Statistical Analysis Plan (2020-08-24): https://cdn.clinicaltrials.gov/large-docs/07/NCT03944707/SAP_000.pdf